CLINICAL TRIAL: NCT04503941
Title: Ultrasound Examination of Inguinal Lymph Node and Knee Joint Slip Fluid Accumulation Was Used to Evaluate the Effect of Acupuncture on Knee Osteoarthritis
Brief Title: Ultrasound Examination of Inguinal Lymph Node Used to Evaluate the Effect of Acupuncture on Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UE of OA
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: A total of 120 patients were enrolled and treated in either the sham-acupuncture (control group) or acupuncture group for 12 weeks, with 8 weeks' follow-up, three times per week.
Who Masked: Participant
Masking Description: Since the acupuncture and sham-acupuncture cannot be blind to the researchers, considering the placebo effect of the subjects, this experiment was blind only to the subjects, namely single-blind. But the researchers did not hint at the treatments received by the patients, and avoided various factors that may have led to bias during the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Experimental): Acupuncture treatment will be the Traditional Chinese Medicine type. Acupuncture 3 times per week, 4 weeks is one treatment period. Every patient will be given 3 treatment period.
  Interventions: Device: Acupuncture treatment
- The control group (Placebo Comparator): False Needle treatment will be the Traditional Chinese Medicine type. Acupuncture 3 times per week, 4 weeks is one treatment period. Every patient will be given 3 treatment period.
  Interventions: Device: False Needle treatment

INTERVENTIONS:
Device: Acupuncture treatment — Acupuncture treatment will be the Traditional Chinese Medicine type. Acupuncture 3 times per week, 4 weeks is one treatment period. Every patient will be given 3 treatment period.
  Arms: Active Comparator
Device: False Needle treatment — False Needle treatment treatment will be the Traditional Chinese Medicine type. Acupuncture 3 times per week, 4 weeks is one treatment period. Every patient will be given 3 treatment period.
  Arms: The control group

SUMMARY:
Knee osteoarthritis (KOA) is a major public health problem among the elderly and is associated with considerable disability. Previous studies on the pathogenesis of this disease mainly focus on cartilage degeneration, but lack of attention to synovitis lesions, and even believe that it is a secondary change in the pathogenesis of osteoarthritis.In recent years, a large number of studies at home and abroad have pointed out that the occurrence and development of knee osteoarthritis are accompanied by synovitis at each stage, and synovial lesions may be the primary manifestation of knee osteoarthritis and affect the evolution of knee osteoarthritis.To this end, some scholars proposed that synovitis lesions as a starting point, may be a new target for the treatment of knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a major public health problem among the elderly and is associated with considerable disability.Under normal circumstances, synovial fluid in the knee joint cavity is absorbed by lymphatic vessels, and the balance of secretion and absorption of synovial fluid in the knee joint is maintained by the lymphatic system.

When there is some kinds of injury of the knee joint synovial received cartilage stimulate, stimulate the synovial vasodilation, synovial cell proliferation activity, produce a large number of joint synovial fluid and secrete a large number of inflammatory liquid, lymphatic metabolism disorder, make joint cavity inflammatory liquid secretion is greater than the absorption, due to the repeated joint fluid absorption and secretion, articular synovial hyperplasia gradually, eventually lost its normal function, a swelling in the knee joint, and the content of inflammatory cytokines in joint fluid, obvious rise, stimulate the immersion in the subchondral bone nerve pain in synovial fluid.In the formation of inflammatory response, the pressure difference between the tissue fluid and the lymphatic vessels promotes the increase of lymphatic reflux, while the input lymphatic vessels tend to converge to the drainage lymph nodes in different regions.Therefore, the observation of changes in lymphatic reflux is more conducive to the evaluation of synovial inflammation and the occurrence of lymph node metastasis. Therefore, regional drainage lymph node metastasis can also be used as an important biological indicator for the evaluation of prognosis and the formulation of treatment strategies.

Acupuncture could be a promising treatment option for knee OA due to the effectiveness of the pain relief and the rarity of adverse effects. In order to get some more reliable data to confirm acupuncture effectiveness on KOA, a long-term follow up interventional study with clear design, standard criteria, control group, will be started to confirm the effects of long term for acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the western medicine diagnostic criteria of knee osteoarthritis;
2. Aged between 50 and 75 years;
3. Patients in line with the 0-III level of radiological classification for knee osteoarthritis degeneration;
4. Patients who did not use glucocorticoid via oral administration or intramuscular, articular, or soft tissue injection four weeks before accepting the test agent;
5. Normal line of force;
6. Patients who signed the informed consent and ensured the compliance.

Exclusion Criteria:

1. Patients with long-term oral administration of agents for knee osteoarthritis, and still in the drug effect period, without elution;
2. Patients with severe heart, brain, liver, kidney or lung dysfunction;
3. Patients with other knee diseases found in arthroscopic surgery;
4. Patients who have accepted other relevant treatments, which may affect the observation on the effects of this study;
5. Patients with mental illness;
6. Patients with coagulation dysfunction;
7. Patients with articular surgical treatment;
8. Patients with a history of abuse of opioid analgesics, sedative hypnotics or alcohol;
9. Patients with poor compliance, who were unable to meet the requirements for follow-up.
10. Pregnant and lactating women.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Ribbens diagnostic criteria | 20 weeks
  Ribbens grading of intra-articular effusion in the ultrasonic knee joint.The thickness of > LMM in the anechoic zone was judged to be joint effusion.
  Classification: level 0: no effusion; level I: small amount of effusion; level II: moderate amount of effusion; level III: large amount of effusion.
Alder blood flow indexing standard | 20 weeks
  Alder blood flow indexing standard for intra-articular effusion in knee joint by ultrasonic Blood flow classification of articular synovium: level 0: no blood flow signal was found in the synovium;Level I: a small amount of blood flow signals can be seen in the synovium, and the blood flow can be seen at points 1-2.Level II: moderate blood flow signal, 1 main blood vessel or 2-3 small blood vessels can be seen at the same time;Class III: rich blood flow, more than 4 blood vessels are visible, or the blood vessels are connected in a network.
Walther standard synovial thickness | 20 weeks
  Walther standard synovium thickness is divided into 4 grades, grade I: thickness <2 mm;Class II: thickness 2-5 mm;Class III: thickness 5-9 mm;Class IV: thickness > 9 mm.
Inguinal lymph node volume | 20 weeks
  Inguinal lymph node
ratio of length to diameter | 20 weeks
  Inguinal lymph node

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Index | 20 weeks
  Western Ontario and McMaster Universities Index for 20 weeks
VAS score | 20 weeks
  VAS score assessed for 20 weeks.
Lequesne index | 20 weeks
  Lequesne index assessed for 20 weeks.
Six-minute walking test | 20 weeks
  Six-minute walking test for 20 weeks.
SF-36 scale | 20 weeks
  Imaging inspection (MRI) assessed for 20 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Ph.D, M.D, Study Director — Shanghai Longhua Hospital
Locations (1):
- Longhua Hospital, Shanghai University of TCM, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
available

REFERENCES:
- [Result] Wang W, Lin X, Xu H, Sun W, Bouta EM, Zuscik MJ, Chen D, Schwarz EM, Xing L. Attenuated Joint Tissue Damage Associated With Improved Synovial Lymphatic Function Following Treatment With Bortezomib in a Mouse Model of Experimental Posttraumatic Osteoarthritis. Arthritis Rheumatol. 2019 Feb;71(2):244-257. doi: 10.1002/art.40696. Epub 2019 Jan 5. PMID 30144298
- [Result] Ribbens C, Andre B, Marcelis S, Kaye O, Mathy L, Bonnet V, Beckers C, Malaise MG. Rheumatoid hand joint synovitis: gray-scale and power Doppler US quantifications following anti-tumor necrosis factor-alpha treatment: pilot study. Radiology. 2003 Nov;229(2):562-9. doi: 10.1148/radiol.2292020206. Epub 2003 Sep 11. PMID 12970463
- [Result] Walther M, Harms H, Krenn V, Radke S, Faehndrich TP, Gohlke F. Correlation of power Doppler sonography with vascularity of the synovial tissue of the knee joint in patients with osteoarthritis and rheumatoid arthritis. Arthritis Rheum. 2001 Feb;44(2):331-8. doi: 10.1002/1529-0131(200102)44:23.0.CO;2-0. PMID 11229463
- [Result] Wauke K, Nagashima M, Ishiwata T, Asano G, Yoshino S. Expression and localization of vascular endothelial growth factor-C in rheumatoid arthritis synovial tissue. J Rheumatol. 2002 Jan;29(1):34-8. PMID 11824968
- [Result] Proulx ST, Kwok E, You Z, Papuga MO, Beck CA, Shealy DJ, Ritchlin CT, Awad HA, Boyce BF, Xing L, Schwarz EM. Longitudinal assessment of synovial, lymph node, and bone volumes in inflammatory arthritis in mice by in vivo magnetic resonance imaging and microfocal computed tomography. Arthritis Rheum. 2007 Dec;56(12):4024-37. doi: 10.1002/art.23128. PMID 18050199
- [Result] Melo Mde O, Pompeo KD, Brodt GA, Baroni BM, da Silva Junior DP, Vaz MA. Effects of neuromuscular electrical stimulation and low-level laser therapy on the muscle architecture and functional capacity in elderly patients with knee osteoarthritis: a randomized controlled trial. Clin Rehabil. 2015 Jun;29(6):570-80. doi: 10.1177/0269215514552082. Epub 2014 Sep 26. PMID 25261425
- [Result] Glimm AM, Werner SG, Burmester GR, Backhaus M, Ohrndorf S. Analysis of distribution and severity of inflammation in patients with osteoarthitis compared to rheumatoid arthritis by ICG-enhanced fluorescence optical imaging and musculoskeletal ultrasound: a pilot study. Ann Rheum Dis. 2016 Mar;75(3):566-70. doi: 10.1136/annrheumdis-2015-207345. Epub 2015 Aug 26. PMID 26311723